CLINICAL TRIAL: NCT01945697
Title: Validation of DNA Methylation Biomarkers for Oral Cancer Detection
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207019
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2014-09

CONDITIONS: Oral Cancer
Keywords: DNA methylation, biomarkers, oral cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cells from oral mouthwash
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal oral mucosa
- oral precancerous lesion or oral cancer

SUMMARY:
The aim of this study is to evaluate the association between several methylated genes and oral cancers. A prospective case control trial is designed with sample size estimated at least 160 cases. It is expected to enroll at least 100 subjects with precancerous lesion or oral cancer, and ~60 subjects with normal oral mucosa. This study is approved by the National Taiwan University Hospital Research Ethics Committee. After signing the informed consent, all of the subjects will receive an intraoral examination and the oral epithelial cells will be collected. If abnormal oral lesion is observed, it will be photographed, and the biopsy will be performed to confirm the diagnosis. For methylated gene detections, the gDNA will be extracted from the collected cells and standardized assay will be performed. Clinical sensitivity and specificity for these methylated genes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age over 20.
* Subject agrees to sign the informed consent form.

Exclusion Criteria:

* Subjects have history of head and neck cancer.
* Subjects have had received chemotherapy for cancers.
* Pregnant Woman
* Subjects whose has oral mucosal lichen planus.
* Subjects whose oral mucosal findings is abnormal, but the diagnosis is unknown.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients come to the Department of Dentistry of National Taiwan University Hospital for oral health care or treatment.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
DNA methylation labeled | 2 years
  To validate the association between the methylation genes and the oral cancer

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Jung Cheng, MD, Principal Investigator — Department of Dentistry National Taiwan University Hospital
Locations (1):
- Department of Dentistry National Taiwan University Hospital, Taipei, Taiwan